CLINICAL TRIAL: NCT06560021
Title: A Randomized Trial of the Utility of Random Biopsies in Patients With Inflammatory Bowel Disease
Brief Title: Utility of Random Biopsies in Patients With Inflammatory Bowel Disease
Acronym: URBI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15225; U01DK138901 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: IBD; UC; inflammatory bowel diseases; colonoscopy; random biopsies; Crohn's disease; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: multicenter parallel group clinical trial
Masking Description: The endoscopist will not be informed of the biopsy strategy until he/she is ready to insert the scope. Participants will not be informed of the randomization until the colonoscopy is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited biopsy strategy (Active Comparator): Targeted biopsies plus 2 random biopsies in 2 segments to assess for inflammation
  Interventions: Other: Biopsy strategy
- Random biopsy strategy (Active Comparator): Targeted biopsies plus 4 biopsies every 10 cm throughout the colon, at a minimum in all segments of the colon known to have been affected by IBD at any time
  Interventions: Other: Biopsy strategy

INTERVENTIONS:
Other: Biopsy strategy — Number of random biopsies, in addition to targeted biopsies, taken during colonoscopies where at least one indication for the colonoscopy is surveillance for dysplasia

SUMMARY:
The proposed study is a multicenter parallel group clinical trial that will include 821 evaluable patients per group who will be randomly assigned to either high definition white light colonoscopy (HDWLC) with targeted biopsies plus 2 random biopsies in 4 segments to assess for inflammation (limited biopsy strategy) or HDWLC with targeted biopsies plus 4 biopsies every 10 cm throughout the colon, at a minimum in all segments of the colon known to have been affected by IBD at any time, regardless of the extent of disease (random biopsy strategy). Participants will be followed until total proctocolectomy or the end of the study period to determine whether the two methods of surveillance colonoscopy are associated with detection of dysplasia or sessile serrated adenoma at follow-up colonoscopy. Follow-up via chart review may continue for up to 15 years from enrollment.

DETAILED DESCRIPTION:
To maximize the yield of surveillance colonoscopy, minimize risk to patients, and deliver cost-effective care, it is imperative to resolve whether random biopsies are warranted for patients with long standing Inflammatory Bowel Disease (IBD) undergoing dysplasia and colorectal cancer (CRC) surveillance with high-definition white light colonoscopy (HDWLC). For this protocol, dysplasia surveillance refers to the process of identifying precancerous dysplasia, sessile serrated adenoma (SSA) or CRC. This protocol describes a pragmatic, multicenter randomized trial of patients with IBD undergoing dysplasia surveillance with HDWLC, the most common type of surveillance colonoscopy performed in the US, to definitively answer this question.

The primary objective of the study is to determine if HDWLC using a limited biopsy strategy is non-inferior to HDWLC using a random biopsy strategy to detect dysplasia or sessile serrated adenoma (SSA) in patients with IBD.

Secondary objectives include:

1. Determine if HDWLC using a limited biopsy strategy is superior to HDWLC with a random biopsy strategy to detect one or more dysplastic or SSA lesion in patients with IBD
2. Determine whether the number of targeted biopsies differs based on the number of random biopsies obtained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of left-sided (greater than 15 cm of disease but not beyond the splenic flexure) or extensive (extending beyond the splenic flexure) ulcerative colitis or IBD-U or colonic Crohn's disease involving at least 1/3 of the colon for at least 8 years
* Patients who are scheduled to undergo colonoscopy as part of routine care.
* At least one indication for the index colonoscopy must be to perform dysplasia surveillance.
* Has not had a colonoscopy in the last 11 months

Exclusion Criteria:

* Any condition that the endoscopist feels is a contraindication to random biopsies
* History of visible (high or low grade) dysplasia not completely removed
* History of sessile serrated adenoma not completely removed
* History of colorectal cancer
* Any condition for which the endoscopist feels that pancolonic contrast or virtual chromoendoscopy is mandatory
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1642 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
number of dysplastic or SSA lesions detected per colonoscopy | At index colonoscopy
  The rationale for this as the primary outcome is that it is important to detect and remove all precancerous lesions. For this outcome, the investigators will include low grade dysplasia (LGD), high grade dysplasia (HGD), SSA or CRC but not indefinite for dysplasia (IFD). Dysplasia will include both conventional and nonconventional forms of dysplasia. Although SSAs do not typically have histologic changes of dysplasia, they are considered precancerous lesions and are more difficult to detect than sporadic adenomatous polyps. The number of dysplastic or SSA lesions will be defined as the number of pathology jars containing a specimen with low-grade or high-grade dysplasia (including CRC) or serrated changes consistent with a sessile serrated adenoma-like change. Even if there are more than one biopsy sample in a jar with dysplasia or SSA, it will be counted as one location with dysplasia or SSA.

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (17):
- United States (17):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - Scripps Health, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Mercy Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF